CLINICAL TRIAL: NCT03541681
Title: A Trial of Repeated Transforaminal Injections With Local Anesthetics With or Without Glucocorticoid in Patients With Cervical Radiculopathy; A Single-center, Randomized Controlled Trial With Short- and Long Term Follow-up
Brief Title: Repeated Transforaminal Anesthetic Injections With or Without Glucocorticoid in Patients With Cervical Radiculopathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study lead could not proceed with the study due to changed employer
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2017/804
Record Dates: First submitted 2018-04-13; First posted 2018-05-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2020-03

CONDITIONS: Neck Pain; Radiculopathy, Cervical; Cervical Foraminal Stenosis; Cervical Disc Disease
Keywords: Epidural Steroid Injections; Cervical Epidural Injections; Transforaminal Epidural Injections; Steroids; Local Anesthetic
MeSH Terms: conditions — Neck Pain; Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoid Injections (Active Comparator): A series of three cervical transforaminal local anesthetic (0,5 ml Bupivacain) injections with glucocorticoid (1 ml Dexamethasone) within 3 months.
  Interventions: Procedure: Glucocorticoid Injections; Procedure: Anesthetic Injections
- Local Anesthetic Injections (Active Comparator): A series of three cervical transforaminal local anesthetic (0,5 ml Bupivacain) injections without glucocorticoid (Dexamethasone) within 3 months.
  Interventions: Procedure: Anesthetic Injections

INTERVENTIONS:
Procedure: Glucocorticoid Injections — 1 ml Dexamethasone + 0,5 ml Bupivacain
  Arms: Glucocorticoid Injections
Procedure: Anesthetic Injections — 0,5 ml Bupivacain

SUMMARY:
The main objective is to evaluate pain and muscle strength in the upper extremities after treatment with cervical transforaminal injection of glucocorticoid vs. transforaminal injection of local anesthetic injection in patients with cervical radiculopathy. The investigators hypothesizes that there are correlations between radiculopathy and muscle weakness.

DETAILED DESCRIPTION:
Previously published studies have not shown a difference in outcome between cervical transforaminal injections with cortisone or local anesthetic in a short term, 6-week, follow-up after using a series of three injections of cervical transforaminal glucocorticoid vs. local anesthetic. No study available thus far has evaluated and compared the long-term effect of these two treatments (glucocorticoid vs. local anesthetics). The investigators aim is to verify if there are responders and non-responders to this type of steroid injections. 100 patients with MRI-verified nerve root compression caused by spondylosis or disc herniation and a history of radiculopathy with or without neck pain and muscle weakness will be included. The participants will be included if they showed at least 50% pain reduction in visual analogue scale (VAS) within 30 min of a diagnostic nerve root block with local anesthetic only. The participants will be blinded and randomized to each treatment group. Pain, muscle weakness, disability and quality of life will be evaluated. Follow-up will be made at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* People >18 years and <65, referred to the department of Neurosurgery in Lund, Sweden for evaluation and treatment of cervical radiculopathy.
* Patients with radiculopathy who after a diagnostic transforaminal injection with 0,5 ml Bupivacain local anesthetics reported a 50% or more reduction of radicular pain according to the visual analogue scale (VAS) (responders).
* Clinical findings and symptoms (i.e. radiculopathy, muscle weakness, sensibility disorder, reflexes) in the upper extremities, correlating to MRI verified nerve root compression on one single level between C4-C7 caused by spondylosis or disc herniation.
* Patients with positive, >50% pain reduction, diagnostic transforaminal injection who choose conservative treatment as first option before surgery.
* Symptoms from dermatome/myotome radiculopathy > 3 months, corresponding to MR-verified foraminal narrowing caused by disc herniation or foraminal stenosis from spondylosis/facet joint hypertrophy.
* Understanding the oral and written consent form in Swedish, and consenting to the study.
* Capable of adhering to the protocol.

Exclusion Criteria:

* Fibromyalgia or other general myalgia not suggestive of radicular pain.
* Cervical myelopathy caused by central spinal stenosis.
* Pain caused by stenosis 3 levels or more and/or disk herniation at 3 levels or more or cervical abnormalities (Klippel-Feil, Lytic/Sclerotic lesions, Recent fractures).
* Previously cervical surgery at the same level or trauma caused by neck distortion i.e. whiplash-associated disorder (WAD).
* Peripheral neuropathy caused by systemic disorders (i.e. diabetes, hereditary, idiopathic or ethanol overconsumption).
* Peripheral nerve compression/entrapment distal to the neuro foramina (i.e. Thoracic outlet syndrome, compression between mm. scalenus, carpal tunnel syndrome)
* Systematic inflammatory diseases involving cervical spine segments and/or spinal cord.
* Neurological motor disorders e.g. ALS and MS.
* Prior medical conditions causing difficulties to participate according to the protocol i.e. stroke, dementia and mental illness.
* Treatment with glucocorticoids injections in the cervical spine within the last 12 months.
* Allergy to glucocorticoid (Dexamethasone) or local anesthetic (Bupivacain).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-06-07 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
VAS - Visual analog scale | 6 months
  VAS evaluates levels of pain intensity using an 10 point scale (range 0-10), with 0 being classified as "no pain", and 10 "worst imaginable pain".

SECONDARY OUTCOMES:
Muscle strength - ISOmetric Power device | 6 months
  Exploratory Outcome Measures
Muscle strength - Commander Echo (JTECH Medical) | 6 months
  Exploratory Outcome Measures
Neck disability index | 6 months
  Neck disability index (NDI), is a patient self-reported questionnaire which contains 10 items including pain, personal care, lifting, reading, headaches, concertation, work, driving, sleeping and recreation. The patient scores each section from 0 to 5. Zero indicates 'no pain' and five indicates 'worst imaginable pain'. The highest possible score of the test is 50 which means complete absence from activity.
EQ-5D-3L | 6 months
  An questionnaire that measures and value changes in health-related quality of life. The 3-level version of EuroQol five Dimensions Questionnaire (EQ-5D-L3) evaluates mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1), some problems (2), and extreme problems (3). The stated value from each dimension converts to a single summary index from 0-1. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
Odom´s criteria | 6 months
  The Odum´s criteria is a patient self-reported evaluation in outcome after degenerative cervical disc surgery. A four graded scale from Excellent (No complaints referable to cervical disc disease; able to continue daily occupation without impairment) to Poor (No improvement, or worse compared with the condition before the operation).
The European Myelopathy Score (EMS) | 6 months
  The European Myelopathy Score (EMS) measures the severity of cervical myelopathy. The questionnaire has five sections divided into different functional criteria, which do not need a baseline or prior examination. Section A evaluates gait and has five levels from "not walking, need wheelchair" to "good gait, climb stairs". Section B evaluates hand function (four levels,) Section C evaluates proprioception and coordination (three levels), Section D evaluates bladder and bowel function (3 levels) and finally Section E evaluates sensory function (3 levels). The maximum sum score for a normal subject is 18 points.

OTHER OUTCOMES:
The Swedish National Spine Register | 6 months
  The Swedish National Spine Register is a patient-based questionnaire. The form contains participants characteristics generic data, VAS, NDI, EMS and EQ-5D and evaluates pre- and postoperative satisfaction with outcome and ability to work.

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Marklund, Professor, Study Director — Region Skane

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Brandt C, Eskilsson A, Tomasevic G. Marklund N. Repeated transforaminal injections in patients with cervical radiculopathy: A randomized trial comparing local anesthetic and glucocorticoid injections on pain and muscle strength. ClinicalTrials.gov [Internet] Identifier Dnr 2017/804, 2018.